CLINICAL TRIAL: NCT01434914
Title: Randomized, Double-blind, Single-center, Placebo-controlled Study to Evaluate the Efficacy of Octenisept® in Patients With Chronic Wounds
Brief Title: Study to Evaluate the Efficacy of Octenisept® in Patients With Chronic Wounds
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: early termination due to poor recruitment
Sponsor: Schülke & Mayr GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OCT-UKE-2011
Record Dates: First submitted 2011-09-13; First posted 2011-09-15 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-05

CONDITIONS: Ulcus Cruris
Keywords: Ulcus cruris; chronic wounds; octenisept®
MeSH Terms: conditions — Foot Ulcer | interventions — octenidine and phenoxyethanol drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- verum (Active Comparator)
  Interventions: Drug: octenisept®
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: octenisept® — Cutaneous solution
  Arms: verum
Drug: Placebo — Cutaneous use
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled trial with octenisept® or placebo in patients with chronic leg ulcers. The study will be conducted at a single center with a total of 70 patients. Patients will be randomized to either the octenisept® group or to the placebo group.

DETAILED DESCRIPTION:
Randomized, double-blind, placebo-controlled trial with octenisept® or placebo in patients with chronic leg ulcers. The study will be conducted at a single center with a total of 70 patients. Patients will be randomized to either the octenisept® group or to the placebo group.

Primary Objectives: Antimicrobial efficacy of octenisept® compared to placebo. Secondary Objectives: Subjective tolerance of octenisept®, evaluation of wound parameters.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients of at least 18 years at the time of consent
* Patients with a venous leg ulcer (Ulcus cruris)
* Patients with a chronic leg ulcer
* Females of childbearing potential who are willing to comply with any applicable contraceptive requirements of the protocol
* Negative pregnancy test
* Satisfactory medical assessment
* Ability to provide written informed consent
* Signed declaration of consent
* Willingness to co-operate

Exclusion Criteria:

* Pregnant or lactating women and women not using contraception
* Known history of alcohol or drug abuse
* Use of any antibiotic medication within the last 7 days prior to the first dose
* Patients with serious concomitant disease
* Patients with a coagulation disorder
* Known history of allergic reactions attributed to octenisept® or one of its compounds
* Participation in another clinical trial within the last 30 days before randomization
* Concomitant treatment with other preparations that interfere with the trial preparation or the disease
* Absence of declaration of consent
* Doubt about willingness to co-operate
* Non-fulfilment of the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2011-10; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Antimicrobial efficacy of octenisept® compared to placebo | 2 weeks after baseline
  Decrease of bacterial load after 2 weeks of treatment

SECONDARY OUTCOMES:
Subjective tolerance of octenisept® | 2 weeks after baseline
  Clinical signs of tolerance of octenisept®
Evaluation of wound parameters | 2 weeks after baseline
  Evaluation of wound healing time and wound size (Planimetry)

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Augustin, MD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany

REFERENCES:
- [Background] Vanscheidt W, Baer M, May TW, Siebert J.: Affecting the wound healing process of chronic ulcera by an octenidine based wound antiseptic. Hyg Med (2005) 30 (5): 153-8
- [Background] Hubner NO, Siebert J, Kramer A. Octenidine dihydrochloride, a modern antiseptic for skin, mucous membranes and wounds. Skin Pharmacol Physiol. 2010;23(5):244-58. doi: 10.1159/000314699. Epub 2010 May 18. PMID 20484966
- See also: Related Info — http://www.schuelke.com